CLINICAL TRIAL: NCT00394225
Title: The Effects of Helium-Hyperoxia on 6-Minute Walking Distance in Chronic Obstructive Pulmonary Disease - A Randomized, Controlled Trial
Brief Title: Helium-Hyperoxia and 6MWT Distance in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BIO-REB 05-186
Record Dates: First submitted 2006-10-30; First posted 2006-10-31 (Estimated); Last update posted 2006-10-31 (Estimated); Status verified 2006-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: 6-Minute Walk Test; COPD; Helium-Hyperoxia; Exercise; Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Oxygen; Helium

INTERVENTIONS:
Drug: Oxygen
Drug: Helium

SUMMARY:
We assessed the effect of altering inspired gas on the 6MWT distance in COPD. We hypothesized that HeO2 would improve walking distance and reduce shortness of breath compared to both RA and O2, and potentially improve quality of life for COPD patients.

DETAILED DESCRIPTION:
We hypothesized that inspiring helium-hyperoxia (HeO2) would significantly improve 6-minute walking test (6MWT) distance in Chronic Obstructive Pulmonary Disease (COPD) subjects.

This was a blinded, randomized crossover study. At Visit 1 we assessed pulmonary function, exercise capacity and 6MWT distance. Visits 2 and 3 consisted of four 6MWT with different inspired gases: room air by mask (RA), 100% O2 by mask (Mask O2), 100% O2 by nasal prongs (Nasal O2), and 70% He/30% O2 by mask (HeO2). Walking distance, shortness of breath, leg fatigue, O2 saturation and heart rate (HR) were assessed

ELIGIBILITY:
Inclusion Criteria:

* Exertional dyspnea
* Activity limitation
* COPD

Exclusion Criteria:

* Recent exacerbation (< 4 wks)
* Supplemental O2
* Significant cardiovascular/musculoskeletal abnormalities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16
Dates: Start 2005-07; Study Completion 2006-05

PRIMARY OUTCOMES:
6 minute walking distance

SECONDARY OUTCOMES:
shortness of breath
leg fatigue
arterial oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Darcy D Marciniuk, MD, FRCP(C), Principal Investigator — University of Saskatchewan
Locations (1):
- Edmonton General Hospital, Caritas Lung HEalth Centre, Edmonton, Alberta, Canada